CLINICAL TRIAL: NCT06928831
Title: The Effect of Flipped Learning and Mobile Teaching Methods on Urinary Catheterization Application Knowledge, Skills and Self-Efficient Level of Nursing Students:Randomized Controlled Trial
Brief Title: The Effect of Teaching Methods on Urinary Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Ozan Konateke
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Nursing Students
Keywords: Nursing students,; Mobile learning,; Flipped learning,; Self-Efficacy,; Urinary Catheterization

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimetal 1 (Experimental): Flipped learning
  Interventions: Other: Experimental
- Experimetal 2 (Experimental): Mobil learning
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — Course materials were shared with the students in the flipped group one week before the theoretical lesson. Google Classroom platform was used so that students could easily access these materials and repeat them at any time and frequency they wanted. A link and QR code were shared with the students to log in to the system. The frequency of downloading and watching the course materials was monitored by the researcher. Next week, the theoretical course was taught in line with the flipped learning model.
  Arms: Experimetal 1
Other: Experimental — The link to the mobile application developed for mobile learning was shared with the students in this group. Students were given 2 weeks to use the application, and students had the opportunity to read and watch the content in the application at any time and frequency they wanted.
  Arms: Experimetal 2

SUMMARY:
Aim: This study was conducted to evaluate the effect of flipped learning and mobile learning methods on nursing students' urinary catheterization application knowledge, skills and self-efficacy level.

Material and Method: The study was conducted as a pretest-posttest randomized controlled experimental research model. It was conducted between June 2023 and April 2025 at Inonu University Faculty of Nursing. The population of the study consisted of all first-year students studying in the department of nursing. The sample consisted of 92 students (Group flipped learning: 30, Group mobile application: 32 and Group control: 30) determined by power analysis. "Individual introduction form", 'Urinary system applications skill evaluation form', 'Knowledge test for urinary system applications' and 'Student self-efficacy scale' were used to collect the data. During the research process, students in the experimental groups were taught with flipped learning and mobile learning methods for two weeks. Students in the control group continued the routine theoretical and practical process.

DETAILED DESCRIPTION:
The Flipped Learning method combines online (prior knowledge acquisition) and face-to-face (learning practices) techniques to offer a learning environment in which the educator takes on a guiding role and the learners are actively engaged in learning experiences. Mobile learning method, on the other hand, provides individualised learning opportunities, enabling students to access educational materials anytime and anywhere and to gain self-managed learning skills. Since this method provides individualised learning opportunities and increases educator-learner interaction, its use in education is becoming increasingly widespread. In this study, both methods were evaluated together and their effects on the development of nursing students' competencies for urinary system practices were evaluated.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or over
* To be enrolled in the 1st year of nursing,
* To receive training on urinary system applications for the first time,
* To have no physical disabilities related to vision, hearing and motor skills,
* To have a smart mobile phone with Android/IOS operating system,
* To volunteer to participate in the study.

Exclusion Criteria:

* Repeating the course,
* Not having a smart mobile phone with Android / IOS operating system,
* Not volunteering to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Efeect of knowledge level | 2 weeks later
  For the pre-test data, 'Individual Introduction Form' and 'Knowledge Test on Urinary System Practices' were given to the students and they were asked to fill them in.
  At the end of 2 weeks, the 'Knowledge Test for Urinary System Practices' was applied again at the end of the 2nd week to see the change in the knowledge levels of the students who were trained with different teaching methods for 2 weeks. There were 25 questions in the knowledge test and 8 experts in the field of nursing were consulted for the questions.
Effect of psychomotor skills | 2 weeks later
  In order to evaluate the psychomotor skill level of the students in the groups, the researcher and the independent observer evaluated the urinary system application skills of each student individually and filled out the 'Urinary System Applications Skill Evaluation Form'. The skill evaluation process of each student lasted 10-15 minutes.
  Skill checklists were developed to evaluate the skill performance of students on urinary system applications. Skill checklists are step-by-step checklists showing the skills expected to be performed by students and were prepared by reviewing the relevant current literature.
Effect of Self-Efficacy | 2 weeks later
  The validity-reliability analysis of the scale developed by Rowbotham and Schmitz to determine the self-efficacy levels of students on nursing students was conducted by Yurtçiçek Eren and Başgöl in 2023. Permission was obtained from the authors for the use of the scale. The scale is four-point Likert-type and has one sub-dimension. The scoring of the scale is '1' Strongly Disagree, '4' Strongly Agree. A score between 10 and 40 can be obtained from the scale, and higher scores indicate an increased sense of self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gulec HY, Aslan H. The effect of conscience perception on job satisfaction and care behaviours in nurses. Arch Psychiatr Nurs. 2024 Jun;50:49-59. doi: 10.1016/j.apnu.2024.03.008. Epub 2024 Mar 11. PMID 38789233